CLINICAL TRIAL: NCT05362968
Title: Strawberries and Risk of Diabetes in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Arpita Basu, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UNLV-2021-252
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: PreDiabetes; Metabolic Syndrome
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Each participants on usual diet and lifestyle for 12 weeks
- Strawberry intervention (Experimental): Each participants will consume freeze-dried strawberry powder (32g/day) for 12 weeks
  Interventions: Drug: Freeze-dried strawberry powder

INTERVENTIONS:
Drug: Freeze-dried strawberry powder — Whole strawberries are freeze-dried to form a powder with improved shelf life that will be used in this research study. Strawberry powder will be provided by the California Strawberry Commission (Watsonville, CA)
  Other Names: Freeze-dried strawberries
  Arms: Strawberry intervention

SUMMARY:
Strawberries can be categorized as a functional food based on results from several clinical trials in improving cardiometabolic health beyond providing nutrition. Recent studies identify the role of strawberries in improving insulin resistance and risks of type 2 diabetes which urgently warrants further investigation, keeping in view the huge public health burden of diabetes in the US. In this study, the investigators propose to investigate the effects of a dietary achievable dose of strawberries on glycemic control, insulin resistance, and HbA1c (primary variables) and biomarkers of inflammation and endothelial function in a 28- week controlled crossover study.

DETAILED DESCRIPTION:
Strawberries are popularly consumed fruits in the US and are a rich source of several bioactive compounds with demonstrated health benefits in T2D and cardiovascular disease (CVD). Based on previously reported studies, strawberries have been shown to improve elevated lipid profiles/dyslipidemia, oxidative stress and inflammation in adults with the metabolic syndrome or prediabetes. In a recently reported study, strawberries at a dose of two-and-a-half servings per day for four weeks was shown to significantly reduce insulin resistance and serum adipokines in obese adults. These results conform to only a few reported trials using strawberries in adults with cardiometabolic risks. While these study findings are clinically meaningful, these warrant urgent investigation in trials of longer duration specifically targeting adults with impaired fasting glucose (vs. other features of the metabolic syndrome) as well as adults with diagnosed T2D with poor glycemic control despite taking medications. Furthermore, to the best of our knowledge, only one clinical trial has been reported on the role of strawberries in improving glycemic control, oxidative stress, and inflammation in adults with T2D. While these results are encouraging, they lack generalizability due to the short duration of the study (six weeks) that precludes accurate changes in glycated hemoglobin (HbA1c) as a stable biomarker of glucose control. Based on these gaps in the existing literature, the investigators will examine the effects of strawberry supplementation at a dose of 2.5 servings/day for 12 weeks on glycemic control and related cardiometabolic profiles in prediabetes in a randomized controlled crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Waist size greater than 40 inches in men or 35 inches in women
* Blood glucose greater than 100mg/dL but less than 126 mg/dL or glycated hemoglobin less than 6.5%
* Insulin resistance >1.0
* Not on diabetes medications
* Normal liver and kidney function tests

Exclusion Criteria:

* Allergy to strawberries
* Smoke or drink alcohol on a regular basis
* Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 12 weeks
  Blood glucose, insulin, glycated hemoglobin
Lipid control | 12 weeks
  Blood total and LDL cholesterol

SECONDARY OUTCOMES:
Inflammation | 12 weeks
  cytokines C-reactive protein adhesion molecules
Diabetes risk hormones | 12 weeks
  adiponectin, leptin
Oxidative stress | 12 weeks
  Serum measures of antioxidants

CONTACTS AND LOCATIONS:
Overall Officials: Arpita Basu, PhD, Principal Investigator — University of Nevada at Las Vegas
Locations (1):
- University of Nevada at Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No